CLINICAL TRIAL: NCT01519011
Title: A PHASE 1, MULTICENTER, OPEN-LABEL STUDY TO EVALUATE THE PHARMACOKINETICS AND EFFECT OF FOOD OF A NEW TABLET FORMULATION OF ORAL AZACITIDINE, AND TO EVALUATE THE SAFETY AND EFFICACY OF ORAL AZACITIDINE IN SUBJECTS WITH MYELODYSPLASTIC SYNDROMES, CHRONIC MYELOMONOCYTIC LEUKEMIA OR ACUTE MYELOID LEUKEMIA
Brief Title: Study to Evaluate Pharmacokinetics, Food Effect, Safety and Efficacy of Oral Azacitidine
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: AZA-MDS-004; T-AZA-006 (Other: Celgene)
Record Dates: First submitted 2012-01-24; First posted 2012-01-26 (Estimated); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute
Keywords: Myelodysplastic Syndromes; MDS; Chronic Myelomonocytic Leukemia; CMML; Acute Myeloid Leukemia; AML; Vidaza; oral azacitidine; aza; oral aza; pharmacokinetics; hematology; myeloid disease; PK
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia, Myelomonocytic, Chronic; Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- 1: A, B, C (Experimental): Dose A: Single oral administration with three 100-mg tablets under fasted condition Dose B: Single oral administration with two 150-mg tablets under fasted condition.
  Dose C: Single oral administration with two 150-mg tablets under fed condition.
  Interventions: Drug: oral azacitidine
- 2: B, C, A (Experimental): Dose A: Single oral administration with three 100-mg tablets under fasted condition Dose B: Single oral administration with two 150-mg tablets under fasted condition.
  Dose C: Single oral administration with two 150-mg tablets under fed condition.
  Interventions: Drug: oral azacitidine
- 3: C, A, B (Experimental): Dose A: Single oral administration with three 100-mg tablets under fasted condition Dose B: Single oral administration with two 150-mg tablets under fasted condition.
  Dose C: Single oral administration with two 150-mg tablets under fed condition.
  Interventions: Drug: oral azacitidine
- 4: B, A, C (Experimental): Dose A: Single oral administration with three 100-mg tablets under fasted condition Dose B: Single oral administration with two 150-mg tablets under fasted condition.
  Dose C: Single oral administration with two 150-mg tablets under fed condition.
  Interventions: Drug: oral azacitidine
- 5: A, C, B (Experimental): Dose A: Single oral administration with three 100-mg tablets under fasted condition Dose B: Single oral administration with two 150-mg tablets under fasted condition.
  Dose C: Single oral administration with two 150-mg tablets under fed condition.
  Interventions: Drug: oral azacitidine
- 6: C, B, A (Experimental): Dose A: Single oral administration with three 100-mg tablets under fasted condition Dose B: Single oral administration with two 150-mg tablets under fasted condition.
  Dose C: Single oral administration with two 150-mg tablets under fed condition.
  Interventions: Drug: oral azacitidine
- Extension (Experimental): 300-mg (three 100-mg tablets) once daily for 21 days of a 28-day cycle.
  Interventions: Drug: oral azacitidine

INTERVENTIONS:
Drug: oral azacitidine — oral azacitidine 300-mg once daily for 3 total doses with two 150-mg tablets (fasted and fed) or three 100-mg tablets (fasted).
  Arms: 1: A, B, C; 2: B, C, A; 3: C, A, B; 4: B, A, C; 5: A, C, B; 6: C, B, A
Drug: oral azacitidine — 300-mg (three 100-mg tablets) once daily for 21 days of a 28-day cycle.
  Arms: Extension

SUMMARY:
The primary purpose of this study is to evaluate the pharmacokinetics of oral azacitidine when administered once daily as two 150-mg tablets, including the effect of food, and to evaluate the bioavailability of oral azacitidine 300-mg when administered as two 150-mg tablets relative to three 100-mg tablets.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of signing the informed consent document
* Diagnosis of Myelodysplastic Syndromes, Chronic Myelomonocytic Leukemia and Acute Myeloid Leukemia
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* At least 3 month life expectancy
* Adequate organ function, defined as:

  * Serum bilirubin ≤ 1.5 times the upper limit of normal (ULN);
  * Serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times the ULN;
  * Serum creatinine ≤ 1.5 times the ULN;
  * Serum bicarbonate ≥ 20 mEq/L
* Females of childbearing potential (FCBP) must:

  * Agree to use at least two effective contraceptive methods (oral, injectable, or implantable hormonal contraceptive; tubal ligation; intra-uterine device; barrier contraceptive with spermicide; or vasectomized partner) throughout the study, and for 3 months following the last dose of oral azacitidine; and
  * Have a negative serum or urine pregnancy test (investigator's discretion; sensitivity of at least 25 mIU/mL) at screening; and
  * Have a negative serum or urine pregnancy test (investigator's discretion; sensitivity of at least 25 mIU/mL) within 72 hours prior to Day 1 of the pharmacokinetic (PK) phase (note that the screening pregnancy test can be used as the test prior to Day 1 of the PK phase if it is performed within the 72 hour timeframe).
* Males with partners who are FCBP must agree that they and their partners will use at least two effective contraceptive methods throughout the study and will avoid fathering a child for 3 months following the date of last oral azacitidine dosing
* Understand and voluntarily sign an informed consent document prior to the start of any study related assessments/procedures
* Able to adhere to the study visit schedule and other protocol requirements

Exclusion Criteria:

* Suspected or proven acute promyelocytic leukemia based on morphology, immunophenotype, molecular assay, or karyotype
* Previous treatment with azacitidine or other demethylating agents within 21 days prior to starting study therapy or ongoing adverse events from previous treatment, regardless of the time period
* Anticancer therapy (standard or investigational) within 21 days prior to starting study therapy or ongoing adverse events from previous treatment, regardless of the time period
* Use of any proton pump inhibitor or any other agent that may affect gastric acid level within 28 days prior to study therapy (only applicable to Part II of the PK phase)
* Concurrent use of erythropoiesis-stimulating agents (ESAs) and other red blood cell hematopoietic growth factors, except that the subject is on a stable dose for at least 4 weeks (28 days) prior to starting study therapy
* Concurrent use of iron-chelating agents, except that the subject is on a stable dose for at least 8 weeks (56 days) prior to starting study therapy
* Concurrent corticosteroid use, except for medical conditions other than Myelodysplastic Syndrome and provided the subject is on a stable or decreasing dose for ≥ 1 week prior to start study therapy
* Pregnant or lactating females
* Any known or suspected hypersensitivity to azacitidine or mannitol or any other ingredient used in the manufacture of oral azacitidine (see the azacitidine IB)
* Uncontrolled systemic fungal, bacterial, or viral infection (defined as ongoing signs/symptoms related to the infection without improvement despite appropriate antibiotics or other treatment)
* Active viral infection with known human immunodeficiency virus (HIV) or viral hepatitis type B or C
* Presence of gastrointestinal disease, malignant hepatic tumors, or other conditions known to interfere with the absorption, distribution, metabolism, or excretion of drugs
* Current congestive heart failure (New York Heart Association Class III-IV Appendix G), unstable angina or angina requiring surgical or medical intervention within 6 months prior to starting study therapy, myocardial infarct within 6 months prior to starting study therapy, or uncontrolled cardiac arrhythmia (defined as arrhythmia that is symptomatic or requires treatment or asymptomatic sustained ventricular tachycardia). Subjects with controlled atrial fibrillation that is asymptomatic are eligible
* Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study
* Any condition that confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-02-07 (Actual); Primary Completion 2012-12-31 (Actual); Study Completion 2015-05-12 (Actual)

PRIMARY OUTCOMES:
PK-(AUC) | Up to 10 days
  PK-Area under the plasma concentration time curve (AUC)
PK-(T½) | Up to 10 days
  PK-Terminal half-life (T½)
PK-(Cmax) | Up to 10 days
  Observed maximum concentration in plasma (Cmax)
PK-(Tmax) | Up to 10 days
  PK-Time to maximum plasma concentration (Tmax)
To evaluate the effect of gastric acid pH modulation, through a proton pump inhibitor, on the PK of oral azacitidine | Up to 10 days
  To evaluate the effect of gastric acid pH modulation, through a proton pump inhibitor, on the PK of oral azacitidine.

SECONDARY OUTCOMES:
Adverse Events | Up to 2 years
  Number of participants with adverse events
Hematological response/improvement | Up to 2 years
  Proportion of subjects achieving hematological response/improvement
Transfusion independence | Up to 2 years
  Proportion of subjects achieving RBC transfusion independence
Platelet transfusion independence | Up to 2 years
  Proportion of subjects achieving platelet transfusion independence

CONTACTS AND LOCATIONS:
Overall Officials: Barry Skikne, M.D., Study Director — Celgene
Locations (8):
- United States (8):
  - Moores UCSD Cancer Center MC-0987, La Jolla, California
  - Rocky Mountain Cancer Center, Denver, Colorado
  - Comprehensive Cancer Centers of Nevada, Las Vegas, Nevada
  - University of Cincinnati Physician's Inc., Cincinnati, Ohio
  - Sarah Cannon Cancer Center, Nashville, Tennessee
  - Texas Oncology, Dallas, Texas
  - Virginia Oncology Associates, Norfolk, Virginia
  - Northwest Cancer Specialists, P.C., Vancouver, Washington

REFERENCES:
- [Background] Laille E, Savona MR, Scott BL, Boyd TE, Dong Q, Skikne B. Pharmacokinetics of different formulations of oral azacitidine (CC-486) and the effect of food and modified gastric pH on pharmacokinetics in subjects with hematologic malignancies. J Clin Pharmacol. 2014 Jun;54(6):630-9. doi: 10.1002/jcph.251. Epub 2014 Jan 18. PMID 24374798
- [Background] Savona MR, Kolibaba K, Conkling P, Kingsley EC, Becerra C, Morris JC, Rifkin RM, Laille E, Kellerman A, Ukrainskyj SM, Dong Q, Skikne BS. Extended dosing with CC-486 (oral azacitidine) in patients with myeloid malignancies. Am J Hematol. 2018 Oct;93(10):1199-1206. doi: 10.1002/ajh.25216. Epub 2018 Sep 3. PMID 30016552